CLINICAL TRIAL: NCT05237115
Title: Helicobacter Pylori Eradication Clostridium Butyricum Capsule and Bacillus Coagulans Tablets With Hydrochloride,Esomeprazole,Amoxicillin and Bismuth-containing Quadruple Therapy: a Randomized,Single-center，Open-label,Phase Ⅳ Trail
Brief Title: Helicobacter Pylori Eradication With Probiotics Combined With Triple Therapy Versus Bismuth-containing Quadruple Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Professor/Chief Physician, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K111111
Record Dates: First submitted 2021-07-12; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Gastritis; Peptic Ulcer; Dyspepsia
Keywords: Helicobacter pylori; Probiotics-combining triple therapy; Bismuth-combining quadruple therapy
MeSH Terms: conditions — Gastritis; Peptic Ulcer; Dyspepsia | interventions — Esomeprazole; Amoxicillin; Clarithromycin; Bismuth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clostridium butyricum group (Experimental): given for 14 days at a dose of Clostridium butyricum capsule 420mg 3 capsules BID, esomeprazole 40 mg BID, amoxicillin 500 mg 2 capsules BID, and clarithromycin 500 mg 1 tablet BID.
  Interventions: Drug: Clostridium butyricum capsule; Drug: esomeprazole; Drug: amoxicillin; Drug: clarithromycin
- Bacillus clotting group (Experimental): given for 14 days at a dose of Bacillus coagulans tablets 350mg 3 capsules BID, esomeprazole 40 mg BID, amoxicillin 500 mg 2 capsules BID, and clarithromycin 500 mg 1 tablet BID.
  Interventions: Drug: esomeprazole; Drug: amoxicillin; Drug: clarithromycin; Drug: Bacillus clotting
- bismuth quadruple therapy (Active Comparator): given for 14 days at a dose of colloidal bismuth tartrate capsule 55 mg 4 capsules BID, esomeprazole 40 mg BID, amoxicillin 500 mg 2 capsules BID, and clarithromycin 500 mg 1 tablet BID.
  Interventions: Drug: esomeprazole; Drug: amoxicillin; Drug: clarithromycin; Drug: Bismuth

INTERVENTIONS:
Drug: Clostridium butyricum capsule — Clostridium butyricum group: given for 14 days at a dose of Clostridium butyricum capsule 420mg 3 capsules BID, esomeprazole 40 mg BID, amoxicillin 500 mg 2 capsules BID, and clarithromycin 500 mg 1 tablet BID.
  Arms: Clostridium butyricum group
Drug: esomeprazole — Esmeprazole 40mg 1tablet BID plus amoxicillin 500 mg 2 capsules BID, clarithromycin 500 mg 1 tablet BID, and colloidal bismuth tartrate capsule 55 mg 4 capsules BID or Bacillus coagulans tablets 350mg 3 capsules BID and Clostridium butyricum capsule 420mg 3 capsules BID as a dose given for bismuth-containing quadruple therapy or probiotics combined with triple therapy.
  Other Names: Nexium
Drug: amoxicillin — Amoxicillin 500 mg 2 capsules BID plus esmeprazole 40mg 1tablet BID, clarithromycin 500 mg 1 tablet BID, and colloidal bismuth tartrate capsule 55 mg 4 capsules BID or Bacillus coagulans tablets 350mg 3 capsules BID and Clostridium butyricum capsule 420mg 3 capsules BID as a dose given for bismuth-containing quadruple therapy or probiotics combined with triple therapy.
  Other Names: Amoxy ( Uni-Amocin )
Drug: clarithromycin — Clarithromycin 500 mg 1 tablet BID plus amoxicillin 500 mg 2 capsules BID, esmeprazole 40mg 1tablet BID, and colloidal bismuth tartrate capsule 55 mg 4 capsules BID or Bacillus coagulans tablets 350mg 3 capsules BID and Clostridium butyricum capsule 420mg 3 capsules BID as a dose given for bismuth-containing quadruple therapy or probiotics combined with triple therapy.
Drug: Bacillus clotting — given for 14 days at a dose of Bacillus coagulans tablets 350mg 3 capsules, esomeprazole 40 mg BID, amoxicillin 500 mg 2 capsules BID, and clarithromycin 500 mg 1 tablet BID.
  Arms: Bacillus clotting group
Drug: Bismuth — given for 14 days at a dose of colloidal bismuth tartrate capsule 55 mg 4 capsules BID, esomeprazole 40 mg BID, amoxicillin 500 mg 2 capsules BID, and clarithromycin 500 mg 1 tablet BID.
  Other Names: Bitnal
  Arms: bismuth quadruple therapy

SUMMARY:
This study aims at evaluating efficacy and safety of probiotics combined with triple therapy (Clostridium butyricum capsule and Bacillus coagulans tablets, esomeprazole, clarithromycin and amoxicillin) versus bismuth-containing quadruple therapy (bismuth,esomeprazole,clarithromycin and amoxicillin) in H. pylori eradication. It is hypothesized that probiotics combined with triple therapy is non-inferior to bismuth-containing quadruple therapy. Patients with confirmed H. pylori positive status will be randomized to one of the treatments described above. At week 2 and 6 follow-up visits, a urea breath test(UBT) will be performed to confirm eradication.

DETAILED DESCRIPTION:
The study will include three phases: screening, treatment and follow-up. Screening: this phase will last a maximum of 28 days and subjects eligibility will be evaluated after informed consent signature. Urea Breath test will be performed in addition to the baseline routine evaluations.

Treatment: Subjects are randomly assigned to treatment and will be treated for 14 days. A randomization visit will take place on Day 0 and an end-of-treatment visit will take place between day 12 and 14.

Follow-up: includes two visits. approximately 14 days of treatment and 28 days after the end of treatment. Eradication of H. Pylori will be confirmed through urea breath test(UBT).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18~75,both gender.
2. Patients with upper gastrointestinal symptoms and with documented H.pylori infection.
3. Patients are willing to receive eradication treatment.
4. Women are eligible if they are not pregnant or nursing, and if they are of childbearing potential they are required to use medically acceptable contraception for the duration of the study and 30 days thereafter.

Exclusion Criteria:

1. Patients are excluded if they have previously used antibiotics to eradicate adequately recorded infection with H. pylori.
2. contraindications or allergies to research drugs.
3. Substantial organ impairment(eg liver cirrhosis, uremia, etc.), severe or unstable cardiopulmonary or endocrine disease.
4. Constant use of anti-ulcer drugs ( including taking proton-pump. inhibitors(PPI) within 2 weeks before the [13C] urea breath test), antibiotics or bismuth complexes (more than 3 times /1 month before screening).
5. Definite diagnosis of gastroduodenal ulcer and MALT's lymphoma.
6. Pregnant or lactating women.
7. Underwent upper gastrointestinal Surgery.
8. highly atypical hyperplasia, have symptom of dysphagia.
9. Evidence of bleeding or iron eficiency anemia.
10. A history of malignancy.
11. Drug or alcohol abuse history in the past 1 year.
12. Systemic use of corticosteroids, non steroidal anti-inflammatory drugs, anticoagulants, platelet aggregation inhibitors (except the use of aspirin for less than 100 mg/d).
13. a person with a mental disorder
14. Enrolled in other clinical trials in the past 3 months.
15. Refusal to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2020-12-05 (Actual); Study Completion 2020-12-05 (Actual)

PRIMARY OUTCOMES:
helicobacter pylori eradication | 28 days after treatment
  The primary end point of this study is H.pylori eradication,established by negative [13C] urea breath test 28 days after the end of eradication.

SECONDARY OUTCOMES:
symptoms effective rates | 14 days of treatment, and 28 days after treatment
  Evaluation effective rate of symptoms 2 weeks of treatment and 4 weeks after the end of treatment.
  Symptom effective rate =（total score before treatment - total score after treatment）/total score before treatment x 100%. Total score = frequency + severity.
  Frequency score is calculated by all the frequency of heartburn,reflux,abdominal pain,and flatulence. Severity is accumulated by the degree of symptoms described above,which is divided to 4 degree as 0 presenting none,and 3 presenting most severe.
adverse events | 14 days of treatment, and 28 days after treatment
  Participants with Adverse Events as a Measure of Safety and Tolerability.The common side effects of the study include headache,dizziness,skin rash,other gastrointestinal disorders,pyrexia,cough and back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Yongquan Shi, Ph. D, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi’an, Shanxi, China